CLINICAL TRIAL: NCT03920111
Title: Flavivirus Cross-priming Potential of Live Attenuated Japanese Encephalitis (JE) Vaccine IMOJEV in Flavivirus naïve and Flavivirus Experienced Participants
Brief Title: Flavivirus Cross-priming Potential of IMOJEV
Acronym: FlaviPrime
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Dr Lance Turtle, Senior Clinical Lecturer, University of Liverpool
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UoL001462 - 4833
Record Dates: First submitted 2019-04-04; First posted 2019-04-18 (Actual); Results first posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - Any status (Other): Up to 3-4 healthy adults
  Interventions: Biological: IMOJEV
- Group 2 - FlaviPrime Naive (Other): Up to 6-8 healthy adults who have never travelled to a flavivirus endemic area and are negative in screening tests for flavivirus immunity.
  Interventions: Biological: IMOJEV
- Group 3 - Flavivirus Exposed (Other): Up to 8-10 healthy adults who have had JE vaccine and/or are previously flavivirus exposed, either through receiving yellow fever vaccine up to 5 years before the study, or from being diagnosed with a flavivirus illness (e.g. dengue or Zika).
  Interventions: Biological: IMOJEV

INTERVENTIONS:
Biological: IMOJEV — live attenuated Japanese encephalitis (JE) vaccine IMOJEV®

SUMMARY:
There is a pressing need for a better experimental system to understand flavivirus antibody responses, beyond dengue, to make sure the investigators are using current vaccines to greatest effect and to inform the development of next-generation vaccines. This study will use live chimeric JE vaccine IMOJEV® as a tool for flavivirus epitope discovery. This will allow experimental JEV infection using replication competent, live, attenuated virus as a model, in a setting where the flavivirus infection history of humans can be tightly controlled.

DETAILED DESCRIPTION:
This study will test the hypothesis that in previously flavivirus-exposed individuals, the antibody response is more broadly cross neutralising, and that this will lead to the identification of conserved virion surface epitopes that could be the target of second generation vaccines.

Exploratory Primary Objectives/Specific aims:

1. To establish a human model system of JEV infection in healthy adult volunteers using live attenuated JE vaccine IMOJEV®.
2. To sort and sequence individual responding B cells (plasmablasts) after vaccination with IMOJEV®, and to generate human monoclonal antibodies to JEV.
3. To generate JEV specific human monoclonal antibodies from the sequences derived in (2).
4. To describe the development, specificity, cross-reactivity and function of the T cell response to IMOJEV®.
5. To establish a sample bank for future work on cross-reactive and other responses to flaviviruses, flavivirus vaccines and other emergent viruses.

Exploratory Secondary Objectives:

1. To examine the specificity and cross-reactivity of the antibody response after JE vaccination, using serum and human monoclonal antibodies.
2. To determine whether there are epitopes which can serve as the target of broadly cross-neutralising antibody responses.

Experimentally the fine specificity and cross-reactivity of the antibody response will be studied by cloning antibodies from plasmablasts (B cells responding to the vaccine) that have been single cell sorted by flow cytometry then sequenced at one week post vaccine. These human monoclonal antibodies will then be mapped on to the surface of the virus particle using established approaches, and tested to look for cross-reactive antibodies. T cell responses to the vaccine will be studied using custom pools of synthetic peptides by ELISpot and flow cytometry.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female adult between 18 and 70 years of age at consent.
2. Written and informed consent obtained from participant and agreement of participant to comply with the requirements of the study
3. Able to attend regularly to donate study blood samples for the duration of the study (8 weeks), no planned re-location or travel to a flavivirus endemic area during the study period.
4. Satisfactory medical screen, as demonstrated by study screening document normal physical examination and normal screening blood tests
5. Group 1: Any flavivirus exposure status; Group 2: No previous flavivirus vaccination (JE, tick borne encephalitis or yellow fever (YF)), no residence in a flavivirus endemic area nor planned travel to a flavivirus endemic area during the period of the study; Group 3: JE vaccine and/or yellow fever vaccine or other proven flavivirus infection within the last 10 years or other proven flavivirus infection (lifetime).
6. An efficacious method of contraception must be used during the study for women of childbearing potential.

Exclusion Criteria:

1. Use of any investigational or non-registered drug within 5 half-lives of the drug, or 30 days preceding administration of study JE vaccine, whichever is longer; or planned use during the study period.
2. Receipt of any investigational biologic agents with mechanisms of action that might affect the immune system, at the discretion of the CI and local PI.
3. Administration of immunosuppressants or other immune-modifying drugs within a period of six months before vaccination or at any time during the study period; participants who have received these agents may also be excluded at the discretion of the CI and local PI.
4. Any confirmed or suspected immunosuppressive or immunodeficient condition.
5. A family history of congenital or hereditary immunodeficiency.
6. Any antiviral drug therapy within a period of 5 drug half-lives or 30 days before vaccination, whichever is longer, or at any time during the study period.
7. History of significant allergic reactions likely to be exacerbated by any component of the study vaccine, especially allergic disease or reactions to any previous dose of any vaccine.
8. History of having received JE vaccine, yellow fever vaccine, tick-borne encephalitis vaccine or experimental flavivirus vaccine (group 2 only).
9. Detectable anti Flavivirus neutralizing antibodies in screening tests (group 2 only).
10. Acute disease (for example acute infection) at the time of enrolment or vaccination, if symptoms are rated as anything more significant than a mild adverse event. Entry into the study and/or vaccination may be deferred until the illness has resolved for at least one week.
11. Acute or chronic, clinically significant in the opinion of the investigator, disease in any organ system, as determined by history, physical examination or laboratory testing.
12. Presence of any inflammatory condition that might require immunomodulatory therapy.
13. Recent blood donation (inclusion can be delayed under these circumstances; the participant should be enrolled 16 weeks after their last blood donation. Each participant should give no more than 470 ml per 16 weeks, so regular blood donation should be suspended during the study and can re-commence 1 month after the last study sample).
14. Current or previous abattoir worker or sheep farmer in Scotland (risk of Louping ill virus exposure; group 2 only).
15. Administration of immunoglobulins and/or any blood products within the three months preceding administration of vaccine, or planned administration during the study period.
16. Seropositive for HIV.
17. Pregnancy or Lactation.
18. History of excessive alcohol consumption (>28 units per week), drug abuse or significant psychiatric illness.
19. Any other condition or consideration that, in the opinion of the Investigator, would pose a health risk to the participant if they were enrolled in the study, or would otherwise interfere with the evaluation of the study aims (e.g. difficult venesection).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lance Turtle, Dr, Principal Investigator — University of Liverpool
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There was difficult in recruiting naïve participants. Therefore the target was changed to 4-8. The total number of participants was not fixed, there was flexibility across the groups, up to a total of 22 participants. The protocol allowed participant replacement if the week 1 blood sample was not collected. This happened to one participant in group 3 who had already received the vaccine, then discontinued. therefore the total number enrolled in this group was 11.
Groups:
- Group 1 - Any Status: Up to 3-4 healthy adults. Participants will be replaced if they withdraw before the one week protocol blood sample.
  IMOJEV: live attenuated Japanese encephalitis (JE) vaccine IMOJEV®
- Group 2 - FlaviPrime Naive: Up to 4-8 healthy adults who have never travelled to a flavivirus endemic area and are negative in screening tests for flavivirus immunity. Participants will be replaced if they withdraw before the one week protocol blood sample.
  IMOJEV: live attenuated Japanese encephalitis (JE) vaccine IMOJEV®
- Group 3 - Flavivirus Exposed: Up to 8-10 healthy adults who have had JE vaccine and/or are previously flavivirus exposed, either through receiving yellow fever vaccine up to 5 years before the study, or from being diagnosed with a flavivirus illness (e.g. dengue or Zika). Participants will be replaced if they withdraw before the one week protocol blood sample..
  IMOJEV: live attenuated Japanese encephalitis (JE) vaccine IMOJEV®
Period: Overall Study
Arm/Group | Group 1 - Any Status | Group 2 - FlaviPrime Naive | Group 3 - Flavivirus Exposed
Started | 4 | 4 | 11
Completed | 4 | 4 | 10 (One participant in group 3 was unable to attend the one week visit, when primary outcome data are collected. This participant was replaced according to the protocol.)
Not Completed | 0 | 0 | 1
Not completed — suspected covid - unable to attend study visit | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Any Status | Group 2 - FlaviPrime Naive | Group 3 - Flavivirus Exposed | Total
Number analyzed (Participants) | 4 | 4 | 11 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 10 | 18
  >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 11
  Male | 1 | 1 | 6 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 3 | 4 | 7 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 4 | 4 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Primary: Plasmablast Percentage of Total B Cells at 7 Days Post Vaccine
Description: Plasmablast percentage of total B cells at 7 days post vaccine Number of plasmablasts sorted by flow cytometry at 7 days post vaccine
Time Frame: 1 week
Population: Percentage of total B cells that are plasmablasts.
Measure: Median (Full Range); unit: percent plasmablasts of B cells
Groups:
- Group 2 - FlaviPrime Naive: Up to 4-8 healthy adults who have never travelled to a flavivirus endemic area and are negative in screening tests for flavivirus immunity.
  IMOJEV: live attenuated Japanese encephalitis (JE) vaccine IMOJEV®
Arm/Group | Group 1 - Any Status | Group 2 - FlaviPrime Naive | Group 3 - Flavivirus Exposed
Number analyzed (Participants) | 4 | 4 | 10
percent plasmablasts of B cells | 1.36 [1.14 to 2.14] | 1.96 [0.98 to 2.65] | 1.69 [0.018 to 3.35]

2. Primary Outcome: Primary: Neutralisation Titre, Measured by 50% of Viral Plaque Reduction at One and Two Months Post Vaccine
Description: Neutralising antibody titre, measured by 50% of viral plaque reduction at one and two months post vaccine
Time Frame: two months
Population: geometric mean +/- 95% confidence interval
Measure: Geometric Mean (95% Confidence Interval); unit: 50% neutralisation titre
Arm/Group | Group 1 - Any Status | Group 2 - FlaviPrime Naive | Group 3 - Flavivirus Exposed
Number analyzed (Participants) | 4 | 4 | 10
50% neutralisation titre
  Antibody titre at 4 weeks post vaccine | 882 [302 to 2574] | 283 [72.7 to 1106] | 932 [568 to 1528]
  Antibody titre at 8 weeks post vaccine | 705 [284 to 1746] | 232 [85.4 to 629] | 931 [554 to 1566]

3. Secondary Outcome: Secondary: Number of Adverse Events Occurring in All Participants in One Month Post Vaccine
Description: Number of adverse events occurring in all participants in one month post vaccine
Time Frame: one month
Measure: Number; unit: Number of adverse events
Arm/Group | Group 1 - Any Status | Group 2 - FlaviPrime Naive | Group 3 - Flavivirus Exposed
Number analyzed (Participants) | 4 | 4 | 11
Number of adverse events | 1 | 0 | 9

ADVERSE EVENTS:
Time Frame: one month post vaccination
Description: Number of adverse events
Arm/Group | Group 1 - Any Status | Group 2 - FlaviPrime Naive | Group 3 - Flavivirus Exposed
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/11
Other Adverse Events (participants affected / at risk) | 1/4 | 0/4 | 6/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Any Status (N=4) | Group 2 - FlaviPrime Naive (N=4) | Group 3 - Flavivirus Exposed (N=11)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Tooth Infection (Infections and infestations) | 0 | 0 | 1 (1)
Parasthesia (Nervous system disorders) | 0 | 0 | 1 (1)
Pulled Right Hamstring (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Right Leg Superficial Thrombophlebitis (Vascular disorders) | 0 | 0 | 1 (1)
Malaise (General disorders) | 0 | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/11/NCT03920111/Prot_000.pdf